CLINICAL TRIAL: NCT02079844
Title: A Randomized, Double-Blind, Placebo Controlled, 3-period, Proof of Mechanism, Cross-Over Study of Roflumilast Administered up to Steady State to Evaluate the Effects of Add-on Roflumilast to Second Generation Antipsychotics on Cognitive Impairment as Well as Brain Imaging (ie, fMRI) and Electrical Activity (ie, EEG) Changes Observed in Subjects With Stable Schizophrenia
Brief Title: Roflumilast Plus Antipsychotics Proof of Mechanism Study in Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ROF-SCHZ_106; 2012-002091-13 (EudraCT Number); U1111-1152-3899 (Other: World Health Organization); 12/SC/0443 (Registry Identifier: NRES)
Record Dates: First submitted 2014-03-04; First posted 2014-03-06 (Estimated); Results first posted 2016-10-03 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-08

CONDITIONS: Schizophrenia
Keywords: Drug therapy
MeSH Terms: conditions — Schizophrenia | interventions — Roflumilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo + Roflumilast 100 μg + Roflumilast 250 μg (Experimental): Roflumilast placebo-matching tablets, orally, once, daily, Days 1 through 8, Period 1, followed by a 14 day washout period, followed by roflumilast 100 μg tablets, orally, once, daily, Days 1 through 8, Period 2, followed by a 14 day washout period, followed by roflumilast 250 μg tablets, orally, once, daily, Days 1 through 8, Period 3. All participants will take a stable dose of second generation antipsychotics throughout the duration of the treatment period.
  Interventions: Drug: Roflumilast; Drug: Placebo; Drug: Second generation antipsychotic
- Roflumilast 100 μg + Roflumilast 250 μg + Placebo (Experimental): Roflumilast 100 μg tablets, orally, once, daily, Days 1 through 8, Period 1, followed by a 14 day washout period, followed by roflumilast 250 μg tablets, orally, once, daily, Days 1 through 8, Period 2, followed by a 14 day washout period, followed by roflumilast placebo-matching tablets, orally, once, daily, Days 1 through 8, Period 3. All participants will take a stable dose of second generation antipsychotics throughout the duration of the treatment period.
  Interventions: Drug: Roflumilast; Drug: Placebo; Drug: Second generation antipsychotic
- Roflumilast 250 μg + Placebo + Roflumilast 100 μg (Experimental): Roflumilast 250 μg tablets, orally, once, daily, Days 1 through 8, Period 1, followed by a 14 day washout period, followed by roflumilast placebo-matching tablets, orally, once, daily, Days 1 through 8, Period 2, followed by a 14 day washout period, followed by roflumilast 100 μg tablets, orally, once, daily, Days 1 through 8, Period 3. All participants will take a stable dose of second generation antipsychotics throughout the duration of the treatment period.
  Interventions: Drug: Roflumilast; Drug: Placebo; Drug: Second generation antipsychotic

INTERVENTIONS:
Drug: Roflumilast — Roflumilast tablets
  Other Names: DALIRESP®; DAXAS®
Drug: Placebo — Roflumilast placebo-matching tablets
Drug: Second generation antipsychotic — Second Generation Antipsychotic (SGA) medication for standard of care therapy will be sourced and managed locally by the site.

SUMMARY:
The purpose of this study is to determine whether cognitive impairment associated with schizophrenia is attenuated by add-on roflumilast administration to second generation antipsychotics (SGA) in participants with stable schizophrenia.

DETAILED DESCRIPTION:
The drug being tested in this study is called roflumilast. Roflumilast is being tested as an add-on treatment to second generation antipsychotics (SGA) to treat cognitive impairment in people with stable schizophrenia. This study will look at improvement in cognitive impairment associated with schizophrenia in people who take roflumilast as an add-on to SGA.

The study will enroll approximately 22 participants. Participants will be randomly assigned (by chance, like flipping a coin) to one of three treatment groups-which will remain undisclosed to the patient and study doctor during the study (unless there is an urgent medical need) All participants will receive the following treatments at different periods throughout the study:

* Roflumilast Dose A + SGA
* Roflumilast Dose B +SGA
* Placebo (dummy inactive pill) - this is a tablet that looks like the study drug but has no active ingredient + SGA.

All participants will be asked to take one tablet at the same time each day throughout the study.

This single-centre trial will be conducted in the United Kingdom. The overall time to participate in this study is up to 64 days. Participants will make 2 screening visits to the clinic and then must be brought to the clinic every day for dosing during each of 3 Treatment Periods. Each Treatment Period will be 8 days in duration. All participants will also make 1 final visit 14 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. Signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Meets schizophrenia criteria as defined by the Diagnostic and Statistical Manual of Mental Disorders (DSM-V) by the Mini International Neuropsychiatric Interview (MINI).
4. On a stable dose of second generation antipsychotics (SGA) for at least 2 months as documented by medical history and assessed by site staff.
5. Meets the following symptom criteria: (a) Positive and Negative Syndrome Scale (PANSS) Conceptual Disorganization item score ≤4 (b) PANSS Hallucinatory Behavior or Unusual Thought Content item scores ≤4 (c) PANSS Negative Subscale scores on all items ≤4.
6. Has cognitive impairment as per investigator judgment.
7. Is aged 18 to 55 years, inclusive, at the time of informed consent.
8. Weighs at least 60 kg and has a body mass index (BMI) between 18 and 32 kg/m^2 inclusive at Screening.
9. A male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 12 weeks after last dose.
10. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to use acceptable methods of contraception from signing of informed consent throughout the duration of the study and for 12 weeks after last dose.
11. Has clinical laboratory evaluations (including clinical chemistry, hematology and complete urinalysis) within the reference range for the testing laboratory, unless the results are deemed not to be clinically significant (NCS) by the investigator at screening and Day 1 of Period 1.

Exclusion Criteria:

1. Has received any investigational compound within 30 days prior to the first dose of study medication.
2. Has received roflumilast in a previous clinical study or as a therapeutic agent.
3. Is an immediate family member, study site employee, or in a dependant relationship with a study site employee who is involved in the conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
4. Has uncontrolled, clinically significant neurological, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, or endocrine disease or other abnormality which may impact the ability of the participant to participate or potentially confound the study results.
5. History of claustrophobia or inability to tolerate mock scanner environment during habituation/screening session.
6. Fulfillment of any of the magnetic resonance imaging (MRI) contraindications on the standard radiography screening questionnaire at the Centre for Neuroimaging Sciences, Institute of Psychiatry, King's College London (ie, history of surgery involving metal implants, metal body piercing, dentures, dental plates or bridges, any implanted device that is electrically, magnetically, and mechanically activated).
7. Has a known hypersensitivity to any component of the formulation of roflumilast.
8. Has a positive urine drug result for drugs of abuse at Screening or Day 1 for each treatment period.
9. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 6 months prior to the screening visit or is unwilling to agree to abstain from alcohol and drugs throughout the study.
10. The participant with a history in the last year or currently receiving treatment with clozapine.
11. Has taken any excluded medication, supplements, or food products.
12. If female, the participant is pregnant or lactating or intending to become pregnant before, during, or within 1 month after participating in this study; or intending to donate ova during such time period.
13. Has evidence of current cardiovascular, hepatic, hematopoietic disease, renal dysfunction, metabolic or endocrine dysfunction, serious allergy, asthma hypoxemia, hypertension, seizures, or allergic skin rash. There is any finding in the participant's medical history, physical examination, or safety laboratory tests giving reasonable suspicion of a disease that would contraindicate taking roflumilast or a similar drug in the same class, or that might interfere with the conduct of the study. This includes, but is not limited to, peptic ulcer disease, seizure disorders, and cardiac arrhythmias.
14. Has current or recent (within 6 months) gastrointestinal disease that would be expected to influence the absorption of drugs (ie, a history of malabsorption, esophageal reflux, peptic ulcer disease, or erosive esophagitis frequent occurrence [more than once per week] of heartburn).
15. History of any surgical intervention known to impact absorption (eg, bariatric surgery or bowel resection).
16. Has a history of cancer within the past 5 years prior to the first dose of study medication. This criterion does not include those participants with basal cell or stage I squamous cell carcinoma of the skin who are eligible.
17. Has a positive test result for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV), human immunodeficiency virus (HIV) antibody/antigen at Screening.
18. Has poor peripheral venous access.
19. Has donated or lost 450 mL or more of his or her blood volume (including plasmapheresis), or had a transfusion of any blood product within 3 months prior to Day 1.
20. Has a Screening or Day 1 of Period 1 abnormal (clinically significant) electrocardiogram (ECG). Entry of any participant with an abnormal (not clinically significant) ECG must be approved, and documented by signature by the principal investigator.
21. Has abnormal Screening or Day 1 of Period 1 laboratory values that suggest a clinically significant underlying disease or participant with the following lab abnormalities: alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >1.5 the upper limits of normal.
22. Has abnormal Screening or Day 1 of Period 1 vital sign values that suggest a clinically significant underlying disease.
23. Has a risk of suicide according to the Investigator's clinical judgment (eg, per Columbia-Suicide Severity Rating Scale [C-SSRS] or has made a suicide attempt within 6 months prior to screening visit).
24. Has a current diagnosis of a significant psychiatric illness other than schizophrenia, per DSM-V and is in an acute phase/episode.
25. In the opinion of the investigator or sponsor, the participant is unsuitable for inclusion in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (1):
- Denmark Hill, London, United Kingdom

REFERENCES:
- [Derived] Gilleen J, Farah Y, Davison C, Kerins S, Valdearenas L, Uz T, Lahu G, Tsai M, Ogrinc F, Reichenberg A, Williams SC, Mehta MA, Shergill SS. An experimental medicine study of the phosphodiesterase-4 inhibitor, roflumilast, on working memory-related brain activity and episodic memory in schizophrenia patients. Psychopharmacology (Berl). 2021 May;238(5):1279-1289. doi: 10.1007/s00213-018-5134-y. Epub 2018 Dec 8. PMID 30536081

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United Kingdom from 13 March 2014 to 15 June 2015.
Pre-assignment Details: Participants with a diagnosis of schizophrenia were enrolled equally in 1 of 3 treatment sequences which determined the order the following 3 treatments were received: placebo, once a day roflumilast 100 μg, roflumilast 250 μg.
Period: Treatment Period 1
Arm/Group | Placebo + Roflumilast 100 μg + Roflumilast 250 μg | Roflumilast 100 μg + Roflumilast 250 μg + Placebo | Roflumilast 250 μg + Placebo + Roflumilast 100 μg
Started | 6 | 7 | 7
Completed | 6 | 7 | 5
Not Completed | 0 | 0 | 2
Not completed — Voluntary Withdrawal | 0 | 0 | 2
Period: Treatment Period 2
Arm/Group | Placebo + Roflumilast 100 μg + Roflumilast 250 μg | Roflumilast 100 μg + Roflumilast 250 μg + Placebo | Roflumilast 250 μg + Placebo + Roflumilast 100 μg
Started | 5 (1 Participant was withdrawn due to an Adverse Event after completing Period 1.) | 7 | 5
Completed | 5 | 6 | 5
Not Completed | 0 | 1 | 0
Not completed — Voluntary Withdrawal | 0 | 1 | 0
Period: Treatment Period 3
Arm/Group | Placebo + Roflumilast 100 μg + Roflumilast 250 μg | Roflumilast 100 μg + Roflumilast 250 μg + Placebo | Roflumilast 250 μg + Placebo + Roflumilast 100 μg
Started | 5 | 5 (1 Participant Voluntarily Withdrew after completing Period 2.) | 5
Completed | 5 | 5 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Roflumilast 100 μg + Roflumilast 250 μg | Roflumilast 100 μg + Roflumilast 250 μg + Placebo | Roflumilast 250 μg + Placebo + Roflumilast 100 μg | Total
Number analyzed (Participants) | 6 | 7 | 7 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.8 (10.13) | 36.9 (10.38) | 48.1 (10.93) | 40.2 (11.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 7
  Male | 4 | 5 | 4 | 13
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 1 | 1 | 2
  Black or African American | 5 | 5 | 4 | 14
  White | 1 | 1 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United Kingdom | 6 | 7 | 7 | 20
Height [Mean (Standard Deviation); unit: cm] | 169.8 (8.68) | 175.0 (7.64) | 169.1 (10.96) | 171.4 (9.14)
Weight [Mean (Standard Deviation); unit: kg] | 79.38 (4.804) | 85.09 (17.406) | 81.41 (15.470) | 82.09 (13.532)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.75 (3.871) | 27.56 (3.823) | 28.20 (3.158) | 27.84 (3.433)
Tobacco Classification [Number; unit: participants]
  Never used tobacco | 1 | 1 | 3 | 5
  Current tobacco user | 2 | 4 | 3 | 9
  Ex-tobacco user | 3 | 2 | 1 | 6
Caffeine Classification [Number; unit: participants]
  Consumes caffeine | 4 | 5 | 5 | 14
  Does not consume caffeine | 2 | 2 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Spatial Span Test Score
Description: The Spatial Span test assesses the participant's working memory. During this task, participants are presented with a board containing blue blocks randomly arranged. The rater first taps out a pattern of blocks, beginning with two blocks and increasing with participant proficiency, and the participant is tasked with tapping the same pattern. After discontinuation of this part of the subtest, the participant is then tasked with tapping out the reverse pattern after the rater's demonstration. These patterns also begin with two blocks and increase with participant proficiency. The total score for this subtest ranges from 0 (worst) to 32 (best). A positive change from Baseline indicates improvement. Analysis of Variance (ANOVA) with treatment sequence, study period, and treatment as fixed effects and participant nested within treatment sequence as a random effect was used for analysis.
Time Frame: Baseline and Day 8 of Treatment Periods 1, 2 and 3
Population: Participants from the Pharmacodynamic Analysis Set, all randomized participants who received at least 1 dose of study drug and had at least 1 pharmacodynamic result post-dose, with data available at both Baseline and Day 8 for analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Placebo: Roflumilast placebo-matching tablets orally, once, daily on Days 1 through 8. All participants took a stable dose of second generation antipsychotics throughout the duration of the treatment period.
- Roflumilast 100 μg: Roflumilast 100 μg tablets, orally, once, daily, Days 1 through 8. All participants took a stable dose of second generation antipsychotics throughout the duration of the treatment period.
- Roflumilast 250 μg: Roflumilast 250 μg tablets, orally, once, daily, Days 1 through 8. All participants took a stable dose of second generation antipsychotics throughout the duration of the treatment period.
Arm/Group | Placebo | Roflumilast 100 μg | Roflumilast 250 μg
Number analyzed (Participants) | 16 | 17 | 16
score on a scale | -0.199 (0.5239) | 0.033 (0.5115) | -0.066 (0.5239)
Statistical Analysis 1: Comparison: Placebo vs Roflumilast 100 μg; Test type: Superiority or Other; p = 0.753, ANOVA — P-values are from ANOVA with treatment sequence, study period, and treatment as fixed effects and subject nested within treatment sequence as a random effect; LS Mean Difference = 0.232, 95% CI 2-sided [-1.269 to 1.733], Standard Error of Mean 0.7313
Statistical Analysis 2: Comparison: Placebo vs Roflumilast 250 μg; Test type: Superiority or Other; p = 0.859, ANOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = 0.133, 95% CI 2-sided [-1.389 to 1.655], Standard Error of Mean 0.7417

2. Primary Outcome: Change From Baseline in Hopkins Verbal Learning Test (HVLT) Score
Description: The HVLT assesses the participant's verbal learning. The test consists of a list of 12 words from three taxonomic categories which are presented orally, and the participant is asked to recall as many as possible after each of three learning trials. The key outcome variable for this task is the total correct responses in the three learning trials. A positive change from Baseline indicates improvement. ANOVA with treatment sequence, study period, and treatment as fixed effects and participant nested within treatment sequence as a random effect was used for analysis.
Time Frame: Baseline and Day 8 of Treatment Periods 1, 2 and 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: correct responses
Arm/Group | Placebo | Roflumilast 100 μg | Roflumilast 250 μg
Number analyzed (Participants) | 16 | 17 | 16
correct responses | -1.699 (1.0813) | 0.239 (1.0617) | 0.677 (1.0829)
Statistical Analysis 1: Comparison: Placebo vs Roflumilast 100 μg; Test type: Superiority or Other; p = 0.131, ANOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = 1.938, 95% CI 2-sided [-0.614 to 4.490], Standard Error of Mean 1.2436
Statistical Analysis 2: Comparison: Placebo vs Roflumilast 250 μg; Test type: Superiority or Other; p = 0.069, ANOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = 2.377, 95% CI 2-sided [-0.198 to 4.951], Standard Error of Mean 1.2545

3. Primary Outcome: Dorsolateral Prefrontal Cortex Activation During the Rewarded Delayed Response Working Memory
Description: BOLD Functional magnetic resonance imaging (fMRI) changes in the blood-oxygen-level-dependent (BOLD) - signal, which changes in response to neural activity. Baseline fMRI measurements will be followed by rewarded delayed response Working Memory (WM) task measurements in which participants are required to remember the spatial location of a target stimulus (a dot) relative to a fixation cross. Participants are given feedback indicating success or failure. ANOVA with treatment sequence, study period, and treatment as fixed effects and participant nested within treatment sequence as a random effect.
Time Frame: Baseline and Day 8 of Treatment Periods 1, 2 and 3
Population: Participants from the Pharmacodynamic Analysis Set, all randomized participants who received at least 1 dose of study drug and had at least 1 pharmacodynamic result post-dose, with data available for analysis.
Measure: Least Squares Mean (Standard Error); unit: unitless parameter estimates
Arm/Group | Placebo | Roflumilast 100 μg | Roflumilast 250 μg
Number analyzed (Participants) | 10 | 10 | 10
unitless parameter estimates | 0.500 (0.1737) | 0.576 (0.1737) | 0.329 (0.1737)
Statistical Analysis 1: Comparison: Placebo vs Roflumilast 100 μg; Test type: Superiority or Other; p = 0.671, ANOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = 0.076, 95% CI 2-sided [-0.739 to 0.106], Standard Error of Mean 0.1757
Statistical Analysis 2: Comparison: Placebo vs Roflumilast 250 μg; Test type: Superiority or Other; p = 0.345, ANOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.171, 95% CI 2-sided [-1.193 to 0.571], Standard Error of Mean 0.1757

4. Secondary Outcome: Change From Baseline in the Continuous Performance Test (CPT)
Description: The CPT is a computerized test that assesses the participant's attention and vigilance. The participant was asked to attend to digits flashing on a computer screen and to click the mouse when the same string of digits flashed consecutively. The test consisted of 3 trials: the first contained 2-digit sequences, the second contained 3-digit sequences, and the third contained 4-digit sequences. Scoring was based the number of correct hits. The total score was an average of the 3 trials. A positive change from Baseline indicates improvement. ANOVA with treatment sequence, study period, and treatment as fixed effects and subject nested within treatment sequence as a random effect was used for analysis.
Time Frame: Baseline and Day 8 of Treatment Periods 1, 2 and 3
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: correct hits
Arm/Group | Placebo | Roflumilast 100 μg | Roflumilast 250 μg
Number analyzed (Participants) | 16 | 17 | 16
correct hits | 0.077 (0.1030) | 0.071 (0.1012) | 0.228 (0.1031)

5. Secondary Outcome: Change From Baseline in Brief Assessment of Cognition in Schizophrenia: Symbol-Coding
Description: The Brief Assessment of Cognition in Schizophrenia (BACS): Symbol-Coding assesses the participant's speed of processing. The test is a timed paper-and-pencil test in which the participant uses a key to write digits that correspond to nonsense symbols. The key outcome variable for this task is the total number of correct, valid symbols in 90 seconds. A positive change from Baseline indicates improvement. ANOVA with treatment sequence, study period and treatment group as fixed effects and participant nested within treatment sequence as a random effect.
Time Frame: Baseline and Day 8 of Treatment Periods 1, 2 and 3
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: correct symbols
Arm/Group | Placebo | Roflumilast 100 μg | Roflumilast 250 μg
Number analyzed (Participants) | 16 | 17 | 16
correct symbols | 0.732 (1.8123) | 0.885 (1.7695) | 2.153 (1.8123)

6. Secondary Outcome: Change From Baseline in Category Fluency Animal Naming Scores
Description: The Category Fluency test assesses the participant's speed of processing. The test is administered orally, with the participant naming as many animals as he can in 1 minute. The key outcome variable for the test is the total number of correct, valid category words in 60 seconds. A positive change from Baseline indicates improvement. ANOVA with treatment sequence, study period, and treatment as fixed effects and participant nested within treatment sequence as a random effect.
Time Frame: Baseline and Day 8 of Treatment Periods 1, 2 and 3
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: correct words
Arm/Group | Placebo | Roflumilast 100 μg | Roflumilast 250 μg
Number analyzed (Participants) | 16 | 17 | 16
correct words | -0.711 (0.8187) | 1.039 (0.8000) | -1.468 (0.8188)

7. Secondary Outcome: Ventrolateral Prefrontal (VLPF) Cortex and Orbitofrontal (OFX) Cortex Activation During the Shift Trials
Description: BOLD fMRI, a test that measures brain activity, was used during the Shifting Task at VLPF and OFX. Participants worked out which pair in a stimulus set consisting of a face and a building; transparent and overlapping, was the target. 1 pair appeared on the left of the screen, the other on the right. In each trial, participants indicated using a button box which side of the screen they thought the target was located on. Every second response, feedback was presented on the screen for 0.6 seconds, indicating whether or not the stimulus chosen was the target. If both of the last 2 choices were correct, the feedback was the word ''correct'' in green; otherwise, the feedback was the word ''incorrect'' in red. After 3 positive feedback events, a change of target occurred. A positive change from Baseline indicates improvement. ANOVA with treatment sequence, study period, and treatment as fixed effects and participant nested within treatment sequence as a random effect was used for analysis.
Time Frame: Baseline and Day 8 of Treatment Periods 1, 2 and 3
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: unitless parameter estimates
Arm/Group | Placebo | Roflumilast 100 μg | Roflumilast 250 μg
Number analyzed (Participants) | 10 | 10 | 10
unitless parameter estimates
  Ventrolateral Prefrontal Cortex (VLPF) | 0.911 (0.3433) | 0.657 (0.3433) | 0.755 (0.3433)
  Orbitofrontal Cortex (OFX) | 0.650 (0.3123) | 0.473 (0.3123) | 0.340 (0.3123)

8. Secondary Outcome: Ventral Striatum Activation During the Reward Trials
Description: BOLD fMRI, a test that measures brain activity, was used during the Reward Task (Monetary Incentive Delay Test). Participants were instructed to respond as quickly as possible to a light-flash on the display screen. The flash was preceded by an arrow icon that informed participants about the consequences of their response to the flash stimulus. Four conditions were included in the paradigm, as follows:
  1. Win condition (arrow up): win 2 pound sterling if the response was sufficiently fast.
  2. Avoidance of loss condition (arrow down: lose 2 pound sterling if the response was too slow.
  3. Verbal control (vertical double arrow): no gain or loss of money.
  4. Passive control condition (horizontal double arrow): No response was required. Each of the above conditions was presented at least 10 times in a random order. ANOVA with treatment sequence, study period, and treatment as fixed effects and participant nested within treatment sequence as a random effect was used for analysis.
Time Frame: Baseline and Day 8 of Treatment Periods 1, 2 and 3
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: unitless parameter estimates
Arm/Group | Placebo | Roflumilast 100 μg | Roflumilast 250 μg
Number analyzed (Participants) | 8 | 8 | 8
unitless parameter estimates | 0.321 (1.0316) | 0.544 (1.0316) | -0.255 (1.0316)

9. Secondary Outcome: Change From Baseline in P300 Amplitude at the Midline Parietal Electrode (Pz)
Description: Brain electrical activity changes were quantified with electroencephalogram (EEG) battery tests. The P300 occurs after the presentation of a novel, behaviorally relevant target stimulus embedded among irrelevant stimuli. It reflects allocation of attention and activation of immediate memory.
  The amplitude of P300 indexes brain actions when the mental representation of the stimulus environment is updated, while its latency indexes stimulus classification speed unrelated to response selection processes. The participants are instructed to push a button when hearing the target stimulus, but not when hearing the standard. They are asked to press the button as fast as possible. A positive change from Baseline indicates improvement. ANOVA with treatment sequence, study period, and treatment as fixed effects and subject nested within treatment sequence as a random effect was used for analysis.
Time Frame: Baseline and Day 8 of Treatment Periods 1, 2 and 3
Population: Participants from the Pharmacodynamic Analysis Set, all randomized participants who received at least 1 dose of study drug and had at least 1 pharmacodynamic result post-dose, with data available for analysis at Baseline and Day 8.
Measure: Least Squares Mean (Standard Error); unit: microvolts (μV)
Arm/Group | Placebo | Roflumilast 100 μg | Roflumilast 250 μg
Number analyzed (Participants) | 16 | 16 | 15
microvolts (μV) | -0.641 (0.9377) | -0.963 (0.9523) | 0.555 (0.9659)

10. Secondary Outcome: Change From Baseline in Mismatch Negativity (MMN) Amplitude at the Midline Frontal Electrode (Fz)
Description: EEG, a test that measures brain electrical activity was performed during the MMN. The MMN is an auditory event related potential that is elicited by any discriminable change in auditory stimulation irrespective of the participant or participant's attention. The response to stimuli is being recorded by EEG electrodes while participants read a book. A positive change from Baseline indicates improvement. ANOVA with treatment sequence, study period, and treatment as fixed effects and subject nested within treatment sequence as a random effect was used for analysis.
Time Frame: Baseline and Day 8 of Treatment Periods 1, 2 and 3
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: μV
Arm/Group | Placebo | Roflumilast 100 μg | Roflumilast 250 μg
Number analyzed (Participants) | 16 | 16 | 15
μV | -0.026 (0.2637) | 0.368 (0.2660) | -0.170 (0.2697)

11. Secondary Outcome: Change From Baseline in Amplitude of the C1 Component of the Visual Evoked Potentials at the Midline Occipital Electrode (Oz)
Description: EEG, a test that measures brain electrical activity was used. Participants had a baseline Visual Evoked Potentials (VEP) recording (2 minute checkerboard VEP) followed by a period of high frequency stimulation (2 minutes 9 Hz checkerboard stimulation). The VEP was repeated 2 minutes after the end of high frequency stimulation. A positive change from Baseline indicates improvement. ANOVA with treatment sequence, study period, and treatment as fixed effects and subject nested within treatment sequence as a random effect was used for analysis.
Time Frame: Baseline and Day 8 of Treatment Periods 1, 2 and 3
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: μV
Arm/Group | Placebo | Roflumilast 100 μg | Roflumilast 250 μg
Number analyzed (Participants) | 16 | 16 | 15
μV | -0.499 (0.6358) | -0.405 (0.6358) | -0.160 (0.6512)

12. Secondary Outcome: Change From Baseline in High Beta/Low Gamma Power During Resting EEG
Description: Participants are asked to open and close their eyes in 30 second alternating blocks to maintain an approximately constant level of arousal. The eyes closed EEG, a test that measures brain electrical activity, is dominated by alpha (8-14Hz) and the eyes open EEG dominated by beta (14-30Hz eyes open) with the two states analyzed separately to increase sensitivity to drug effects in these bands. Ratio is calculated as High Beta/Low Gamma Power. A positive change from Baseline indicates improvement. ANOVA with treatment sequence, study period, and treatment as fixed effects and subject nested within treatment sequence as a random effect.
Time Frame: Baseline and Day 8 of Treatment Periods 1, 2 and 3
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Placebo | Roflumilast 100 μg | Roflumilast 250 μg
Number analyzed (Participants) | 16 | 17 | 15
ratio | -0.127 (0.0689) | -0.078 (0.0673) | -0.040 (0.0709)

13. Secondary Outcome: Change From Baseline in Frontal Theta Power (EEG) During N-Back Working Memory Task
Description: EEG, a test that measures brain electrical activity, was performed during the n-back task. In the n-back task participants are required to monitor a series of letters and report when the current letter matches the letter n integers back, where n=1 (1-back) or n=2 (2-back), the latter requiring a greater working memory resources. The task requires continuous updating of information stores. In the 0-back condition (which does not require manipulation of material in working memory), participants respond to the appearance of a pre-specified letter. The task consists of alternating 30-second (s) blocks of 0-back with 1-back, and 2-back conditions, with letters displayed every 2 s for 1 s within each block. A positive change from Baseline indicates improvement. ANOVA with treatment sequence, study period, and treatment as fixed effects and subject nested within treatment sequence as a random effect was used for analysis.
Time Frame: Baseline and Day 8 of Treatment Periods 1, 2 and 3
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: μV
Arm/Group | Placebo | Roflumilast 100 μg | Roflumilast 250 μg
Number analyzed (Participants) | 16 | 16 | 15
μV | -0.068 (0.0482) | -0.073 (0.0490) | 0.002 (0.0497)

14. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score
Description: PANSS assesses the positive symptoms, negative symptoms, and general psychopathology associated with schizophrenia. The scale consists of 30 items. Each item is rated on a scale from 1 (symptom not present) to 7 (symptoms extremely severe). Positive subscale consists of 7 items which assesses the positive symptoms with subscale score ranging from 7 to 49, where higher score indicates greater severity. Negative subscale consists of 7 items which assesses the negative symptoms with subscale score ranging from 7 to 49, where higher score indicates greater severity. General psychopathology subscale consists of 16 items which assesses the general symptoms of schizophrenia with subscale score ranging from 16 to 96, where higher score indicates greater severity. A negative change from Baseline indicates improvement. ANOVA with treatment sequence, study period and treatment group as fixed effects and participant nested within treatment sequence as a random effect was used for analysis.
Time Frame: Baseline and Day 8 of Treatment Periods 1, 2 and 3
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Roflumilast 100 μg | Roflumilast 250 μg
Number analyzed (Participants) | 16 | 17 | 15
score on a scale
  Total Positive Score | -0.737 (0.9939) | -0.670 (0.9821) | -0.196 (1.0098)
  Total Negative Score | 1.480 (1.0653) | 1.580 (1.0484) | 0.650 (1.0876)
  Total General Psychopathology Score | 0.313 (1.5978) | -1.457 (1.5700) | -0.959 (1.6344)

15. Secondary Outcome: Percentage of Participants Who Experience at Least 1 Treatment-Emergent Adverse Event
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: From Day 1 until Day 63
Population: Safety population included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Roflumilast 100 μg | Roflumilast 250 μg
Number analyzed (Participants) | 16 | 17 | 19
percentage of participants | 56.3 | 41.2 | 47.4

16. Secondary Outcome: Percentage of Participants Who Meet the Markedly Abnormal Criteria for Safety Laboratory Tests
Description: Percentage of participants with markedly abnormal safety laboratory tests (Hematology, Serum Chemistry and Urinalysis) collected throughout the study.
Time Frame: From Day 1 until Day 63
Population: Safety population, including all randomized participants who received at least 1 dose of study drug and completed the laboratory tests during treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Roflumilast 100 μg + Roflumilast 250 μg | Roflumilast 100 μg + Roflumilast 250 μg + Placebo | Roflumilast 250 μg + Placebo + Roflumilast 100 μg
Number analyzed (Participants) | 5 | 7 | 5
percentage of participants
  Hematology | 0 | 0 | 20.0
  Serum Chemistry | 20.0 | 14.3 | 0
  Urinalysis | 0 | 0 | 0

17. Secondary Outcome: Percentage of Participants Who Meet the Markedly Abnormal Criteria for Vital Sign Measurement
Description: Vital signs were oral body temperature, respiration rate, supine blood pressure (after 5 minutes resting), and pulse rate.
Time Frame: From Day 1 until Day 63
Population: Safety population, including all randomized participants who received at least 1 dose of study drug and completed the vital sign tests on Day 8 of each treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Roflumilast 100 μg | Roflumilast 250 μg
Number analyzed (Participants) | 16 | 17 | 16
percentage of participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 63 Days
Description: At each visit the investigator had to document any occurrence of adverse events and clinically significant abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | Roflumilast 100 μg | Roflumilast 250 μg
Serious Adverse Events (participants affected / at risk) | 1/16 | 0/17 | 0/19
Other Adverse Events (participants affected / at risk) | 8/16 | 7/17 | 9/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=16) | Roflumilast 100 μg (N=17) | Roflumilast 250 μg (N=19)
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=16) | Roflumilast 100 μg (N=17) | Roflumilast 250 μg (N=19)
Palpitations (Cardiac disorders) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Gingival swelling (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Catheter site bruise (General disorders) | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 2 | 1
Beta haemolytic streptococcal infection (Infections and infestations) | 0 | 0 | 1
Tinea pedis (Infections and infestations) | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 1 | 2
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Middle insomnia (Psychiatric disorders) | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Scar pain (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.